CLINICAL TRIAL: NCT05378672
Title: Phase 3, Single-administration, Open-label Trial to Assess the Efficacy, Safety, PK, and PD of Dasiglucagon When Administered as a Rescue Therapy for Severe Hypoglycemia in Pediatric Patients Below 6 Years of Age With Type 1 Diabetes (T1D)
Brief Title: A Study to Inv. Safety, Efficacy & PD of Dasiglucagon as Hypoglycemia Rescue Therapy in Children <6 Years With T1D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP4207-21052
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hypoglycemia; Type 1 Diabetes
Keywords: Hypoglycemia; Low Blood Sugar; Type 1 Diabetes; Diabetes; T1D
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — dasiglucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dasiglucagon 0.6 mg (Experimental): Participants will receive a single dose of 0.6 mg dasiglucagon.
  Interventions: Drug: Dasiglucagon
- Dasiglucagon 0.3 mg (Experimental): Participants will receive a single dose of 0.3 mg dasiglucagon.
  Interventions: Drug: Dasiglucagon

INTERVENTIONS:
Drug: Dasiglucagon — Dasiglucagon, 0.6 mg/0.6 mL or 0.3 mg/0.3 mL will be administered as an under the skin (subcutaneous, s.c.) injection by a prefilled syringe, into the buttocks.
  Other Names: Zegalogue, ZP4207

SUMMARY:
This research study will investigate whether dasiglucagon as a rescue therapy for participants under 6 years of age works and is safe to use. In addition, the study will investigate how dasiglucagon works in the body (pharmacokinetics and pharmacodynamics).

Participants will receive 1 single dose as an injection under the skin (subcutaneous, s.c.) into the buttocks.

Participants will have 3 visits with the study team. For each participant, the study will last up to 84 days.

DETAILED DESCRIPTION:
This trial will use a single-administration, open-label trial design to assess the ability of a single SC injection of dasiglucagon to increase plasma glucose in pediatric children with T1D with hypoglycemia. A total of 8 children will be included; 4 children receiving a dose of 0.3 mg and 4 children receiving a dose of 0.6 mg. Of the 4 children receiving 0.3 mg, 2 children should preferably be below 2 years at screening. The 2 additional children receiving 0.3 mg should weigh below 15 kg at screening and should preferably be below 4 years at screening. For children receiving the 0.6 mg dose, all must be above 2 years at screening. Before an eligible child is dosed, the dose level (0.6 mg or 0.3 mg) must be confirmed by the sponsor. Each child will be dosed after the safety assessment of the preceding child has been completed and assessed by the Trial Safety Group.

The trial will include the following visits:

* A screening visit (Visit 1) in the period from Day - 50 to Day - 29 (pre-treatment visit)
* A dosing visit (Visit 2), Day 1 (day of single dosing with investigational medicinal product [IMP])
* A Safety follow-up visit (Visit 3) at Day 29 +5 days (the end-of-trial visit).

The primary endpoint of the trial is plasma glucose change from baseline at 30 minutes after IMP injection or at the time of rescue by intravenous glucose. Pharmacodynamics (PD) i.e., plasma glucose will be assessed at baseline and 15 and 30 minutes after dosing, while the glucose levels will be monitored by continuous glucose monitoring and by a plasma glucose analyzer during the dosing visit (Visit 2). Pharmacokinetics (PK) will be assessed throughout a 300-minute period at the dosing visit (Visit 2). Safety will be assessed prior to dosing and throughout a 300-minute period after dosing and again at the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are confirmed as having T1D based on medical history and are receiving daily insulin therapy via insulin pump or MDI
* Body weight greater than 8 kg
* Child must be <6 years of age at the time of screening
* Further inclusion criteria apply

Exclusion Criteria:

* Known or suspected allergy to the IMP or related products
* Any condition that in the investigators opinion may result in diminished hepatic glycogen stores (e.g., prolonged fasting (more than 24 hours) at Visit 2
* History of anaphylaxis or symptoms of severe systemic allergy (such as angioedema)
* History of hypoglycemic events associated with seizures
* Further exclusion criteria apply

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Zealand Pharma A/S
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cook Childrens Health Care System, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the United States.
Pre-assignment Details: A total 10 participants were screened of which 2 were screen failures and 8 were enrolled to receive study treatment.
Groups:
- Dasiglucagon 0.3 mg: Participants received a single dose of 0.3 milligrams (mg) dasiglucagon subcutaneous (SC) injection on Day 1.
- Dasiglucagon 0.6 mg: Participants received a single dose of 0.6 mg dasiglucagon SC injection on Day 1.
Period: Overall Study
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants who were enrolled and received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Dasiglucagon 0.3 mg: Participants received a single dose of 0.3 mg dasiglucagon SC injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.5 (1.00) | 4.0 (0.82) | 3.3 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Glucose Concentration at 30 Minutes After IMP Injection
Description: Glucose levels were monitored by continuous glucose monitoring and by a plasma glucose analyzer.
Time Frame: Baseline, 30 minutes after dosing on Day 1
Population: Full analysis set (FAS) included all participants of the SAF. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 4 | 3
milligrams per deciliter (mg/dL) | 102.3 (10.72) | 104.3 (14.47)

2. Secondary Outcome: Change From Baseline in Plasma Glucose Concentration at 15 Minutes After IMP Injection
Description: Glucose levels were monitored by continuous glucose monitoring and by a plasma glucose analyzer.
Time Frame: Baseline, 15 minutes after dosing on Day 1
Population: FAS included all participants of the SAF. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 4 | 3
mg/dL | 57.3 (13.84) | 53.3 (4.04)

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergence was defined as those adverse events (AEs) that occurred after dosing and those existing AEs that worsened during the study. An AE was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the trial intervention.
Time Frame: From first dose of study drug up to end of follow up (up to Day 29)
Population: SAF included all participants who were enrolled and received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 4 | 4
Participants | 3 | 4

4. Secondary Outcome: Number of Participants Who Received Rescue Intravenous (IV) Glucose Infusion Administration
Time Frame: Within 30 minutes of infusion on Day 1
Population: SAF included all participants who were enrolled and received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

5. Secondary Outcome: Time to First IV Glucose Infusion Following Treatment With Dasiglucagon
Description: Time to first IV glucose infusion (minutes) was defined as Time of start of first glucose administration - Time of administration of study medication.
Time Frame: Start of first glucose administration up to 30 minutes post-infusion on Day 1
Population: SAF included all participants who were enrolled and received at least 1 dose of IMP. Here, "Overall Number of Participants Analyzed" is '0' because no participants received glucose infusion.
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of follow up (up to Day 29)
Arm/Group | Dasiglucagon 0.3 mg | Dasiglucagon 0.6 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon 0.3 mg (N=4) | Dasiglucagon 0.6 mg (N=4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon 0.3 mg (N=4) | Dasiglucagon 0.6 mg (N=4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Application site rash (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT05378672/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT05378672/SAP_001.pdf